CLINICAL TRIAL: NCT03149887
Title: Use of Liposomal Bupivacaine for Postoperative Pain Management After Arthroscopic Rotator Cuff Repair
Brief Title: Liposomal Bupivacaine After Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steven Orebaugh (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor-Investigator, Steven Orebaugh, Professor of Anesthesiology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PRO17020089
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Results first posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Injection of liposomal bupivacaine in surgical field at end of arthroscopic rotator cuff repair.
  Interventions: Drug: Liposomal bupivacaine
- Control (Active Comparator): Injection of inert placebo solution in surgical field at end of arthroscopic rotator cuff repair.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liposomal bupivacaine — Liposomal bupivacaine solution (Exparel) for injection
  Other Names: Exparel
  Arms: Experimental
Drug: Placebo — Inert solution created to appear as liposomal bupivacaine (Exparel) for injection
  Other Names: Placebo solution for liposomal bupivacaine (Exparel)
  Arms: Control

SUMMARY:
Liposomal bupivacaine, a long-acting form of bupivacaine, has been found to be effective for postoperative pain control after total knee, total hip and total shoulder arthroplasty. We are conducting a randomized, controlled trial to evaluate pain control after arthroscopic rotator cuff repair in ambulatory patients, comparing standard care in the control group, with standard care plus the addition of injection of liposomal bupivacaine in the experimental group.

DETAILED DESCRIPTION:
Arthroscopic rotator cuff repair is among the most painful of orthopedic surgeries (1-3). Hundreds of thousands of these procedures are carried out in the U.S. each year. Many involve the use of a brachial plexus nerve block, which serves to control pain for 12 to 14 hours. However, when the block wears off, many patients are left with severe pain. (4-5) This severe pain must then be managed at home with oral opioids, which have numerous undesirable side effects, and may lead to chronic opioid dependence. Thus, any therapy which might reduce the pain burden on these patients and therefore reduce opioid use and side effects, would be advantageous.

Recently, a long-acting form of bupivacaine, prepared in liposomes, has been approved for use by injection in the surgical field, though not for peripheral nerve blockade (6). The drug has been used to improve postoperative pain after total knee arthroplasty and total hip arthroplasty when injected in the peri-articular tissues by the orthopedist (7-12), as well as in other surgeries, both orthopedic and non-orthopedic.(13-16) Unfortunately, preliminary studies utilizing liposomal bupivacaine as the injectate in peripheral nerve blocks have been disappointing, largely because the gradual release of the drug did not permit establishment of effective nerve blockade; it appears to be more effective in the role of analgesic as opposed to anesthetic (17).

In addition to lower extremity orthopedic procedures, liposomal bupivacaine has also been demonstrated to reduce pain after shoulder arthroplasty (joint replacement), a similarly painful shoulder procedure. Liposomal bupivacaine is FDA approved for administration into surgical sites to produce postsurgical analgesia and mitigate pain, but it hasn't been evaluated yet as an intervention to provide analgesia for rotator cuff surgery, though the pain mechanisms for these two procedures, including joint capsule violation and boney intervention are likely similar.

In this prospective, comparative, randomized, double blinded, placebo controlled trial, we propose to provide standard therapy for both groups of patients, consisting of interscalene block with 16 ml of standard 0.5% bupivacaine, as well as propofol infusion to provide general anesthesia in the operating room and low doses of ketamine for analgesia. In addition, half of the patients will receive an injection of 266 mg liposomal bupivacaine (FDA approved dosage) into the subacromial space and peri-articular tissues at the end of surgery. The other half of the patients will receive an injection of an inert solution of comparable volume into the peri-articular tissues at the conclusion of surgery (control group).

The primary outcome measure is pain score at the time of block resolution, as noted by patients when called at 24 hours after surgery. Secondary outcomes include maximal pain score on postoperative day 1, 2 and 3, total oral opioid morphine equivalent after 3 days, and occurrence of typical opioid side effects (nausea, vomiting, drowsiness). In addition to follow up phone call on postoperative day 1, patients will keep a pain diary, documenting pain scores and opioid use for the first 72 hours, which will be collected by the surgeon in his office at the first postoperative visit. Any adverse occurrences related to nerve blockade or prolonged bupivacaine effect will also be recorded.

We expect to enroll 25 patients in each group (total of 50). Sample size is based upon the a priori assumption that liposomal bupivacaine will result in reduced pain scores by at least 2 units on the NRS scale at the time of nerve block resolution. Inclusion criteria include adult patients, undergoing rotator cuff repair as outpatients at our facility, ASA physical status category 1 through 3. Exclusion criteria include inability to receive local anesthetic medications for any reason, contraindications to peripheral nerve block (coagulopathy, patient refusal, local infection and pre-existing nerve injury or dysfunction in the operative arm), chronic opioid dependence, pregnancy and pediatric age group. This study will involve anesthesiology, orthopedics, physical therapy, pain management and the center for translational science institute at the University of Pittsburgh.

References:

1. Kim CW, Kim JH, Kim DG. The factors affecting pain pattern after arthroscopic rotator cuff repair. Clin Orthop Surg. 2014;6:392-400.
2. Uquillas CA, Capogna BM, Rossy WH, Mahure SA, Rokito AS. Post operative pain control after arthrosopic rotator cuff repair. Review JSES 2016.25(7): 1204-13.
3. Shin SJ, Do NH, Lee J, Ko YW. Efficacy of a subacromial corticosteroid injection for persistent pain after arthroscopic rotator cuff repair. Am J Sports Med 2016. 44(9):2231-6.
4. Abdallah FW, Halpern SH, Aoyama K, Brull R. Will the real benefits of single-shot interscalene block please stand up? A systematic review and meta-analysis. Anesth Analg. 2015. 120(5):1114-29.
5. Mifune Y, Inui A, Nagura I, Sakata R, Muto T, Harada Y, TAkase F, Kurosaka M, Kokubu T. Application of pain quantitative analysis device for assessment of post operative pain after arthroscopic rotator cuff repair. Open Orthoped J. 2015.9:89-93.
6. Ilfeld BM. Liposome bupivacaine in peripheral nerve blocks and epidural injections to manage postoperative pain. Exp Opin Pharm. 2013. 14(17):2421-31.
7. Iorio R. The role of liposomal bupivacaine in vale-based care. Am J Ortho. 2016. 45(7):S13-S17.
8. Sporer SM, Rogers T. Postoperative pain management after primary total knee arthroplasty: The value of liposomal bupivacaine. J Arthroplasty. 2016. 31(11):2603-2607.
9. Chugtai M, Cherian JJ, Mistry JB, Elmallah RD, Bennett A, Mont MA. Liposomal bpuivicaine suspension can reduce lengths of stay and improve discharge status of patients undergoing total knee arthroplasty. J Knee Surg. 2016. 29(5):e3
10. Yu SW, Szulc AL, Walton SL, Davidovitch RI, Bosco JA, Iorio R. Liposomal bupivacaine as an adjunct to postoperative pain control in total hip arthroplasty. J Arthroplasty. 2016. 31(7):1510-5.
11. Cien AJ, Penny PC, Horn BJ, Popovich JM, Taunt CJ. Comparison between liposomal bupivicane and femoral nerve block in patients undergoing primary total knee arthroplasty. J Surg Orthop Adv. 2015. 24(4):225-9.
12. Barrington JW, Olugbode O, Lovald S, Ong K, Watson H, Emerson RJ. Liposomal bupivacaine: A comparative study of more than 1000 total joint arthroplasty cases. Orthoped Clin Na. 2015. 46(4):469-77.
13. Robbins J. Green CL. Parekh SG. Liposomal bupivacaine in forefoot surgery. Foot Ankle Int. 2015. 36(5):503-7.
14. Huh J, Parekh SG. Liposomal bupivacaine in hallux valgus surgery: a multimodal pain management adjunct. J Surg Orthop Adv.2014. 23(4):198-202.
15. Hutchins JL, Kesha R, Blanco F, Dunn T, Hochhalter R. Ultrasound-guided subcostal transversus abdominus plane blocks with liposomal bupivacaine vs. non-liposomal bupivacaine for posteropative pain control after laparoscopic hand-assisted donor nephrectomy: a prospective randomized observer-blinded study. Anaesthesia. 2016. 71(7):930-7.
16. Miranda SG, Liu Y, Morrison SD, Sood RF, Gallagher T, Gougoutas AJ, Colohan SM, Loui O, Mathes DW, Neligan PC, Said HK. Improved health care economic outcomes after liposomal bupivacaine administration in first-stage breast reconstruction. J Plast Reconstr Aesthet Surg. 2016. 69(10):1456-7.
17. Ilfeld BM, Malhotra N <Furnish TJ, Donohue MC, Madison SJ. Liposomal bupivacaine as a single injection peripheral nerve block: a dose-response study. Anesth Analg.2013. 117(5):1248-56.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients up to age 65 years, undergoing elective, ambulatory, arthroscopic rotator cuff repair.

Exclusion Criteria:

* Pregnancy, coagulopathy, allergy to bupivacaine, renal failure, hepatic insufficiency, and/or inappropriate candidate for usual therapy (specifically, if unable to receive the usual preoperative interscalene nerve block: preexisting nerve injury on side of surgery, refusal of nerve block, infection at site of nerve block).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center-Southside/Mercy, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 54 patients recruited at time of presentation for surgery. These 54 received the injection of either liposomal bupivacaine (experimental group) or normal saline (control group).
Groups:
- Experimental (Liposomal Bupivacaine): Injection of liposomal bupivacaine in surgical field at end of arthroscopic rotator cuff repair.
  Liposomal bupivacaine: Liposomal bupivacaine solution (Exparel) for injection
- Control (Normal Saline): Injection of Placebo solution in surgical field at end of arthroscopic rotator cuff repair.
  Placebo: Normal saline in same volume as exparel injection in experimental group
Period: Overall Study
Arm/Group | Experimental (Liposomal Bupivacaine) | Control (Normal Saline)
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control (Normal Saline): Injection of normal saline in surgical field at end of arthroscopic rotator cuff repair.
  Placebo: Normal saline in volume equal to that of the liposomal bupivacine injected in experimental group
- Total: Total of all reporting groups
Arm/Group | Experimental (Liposomal Bupivacaine) | Control (Normal Saline) | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (7.2) | 56.3 (7.8) | 57.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 14 | 14 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Pain Score [NRS] at Time of Block Resolution
Description: Numeric rating score pain level at time of nerve block resolution, on scale of 0-10, as reported by patient at time of 24 hour follow up phone call. A reported score of zero implies no pain, whereas a score of "10" implies very severe pain. Outcome score is mean of reported pain scores by participants at time of nerve block resolution.
Time Frame: At the time of block resolution, as reported by patients at follow up phone call
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Control (Normal Saline): Injection of saline solution in surgical field at end of arthroscopic rotator cuff repair.
  Placebo: Saline solution injected in surgical field in same volume as liposomal bupivacaine injected in experimental group.
Arm/Group | Experimental (Liposomal Bupivacaine) | Control (Normal Saline)
Number analyzed (Participants) | 27 | 27
Score on a scale | 5.4 (2.6) | 5.8 (3.2)
Statistical Analysis 1: Comparison: Experimental (Liposomal Bupivacaine) vs Control (Normal Saline); Test type: Superiority; p = 0.66, t-test, 2 sided

2. Secondary Outcome: Mean NRS Pain Score at Rest on Postoperative Day 1
Description: Mean NRS pain score on scale of 1-10, at rest (zero is no pain, 10 is severe pain). Patients recorded their pain score at rest with administration of each oral analgesic tablet. Outcome score is mean of reported pain scores for this day.
Time Frame: Postoperative day 1
Population: These 51 patients underwent the injection, were assessed for the primary outcome, and completed the questionnaire related to the pain, analgesic and side effects for first three postoperative days (secondary outcomes). Three patients did not fill out this questionnaire and therefore are not included in the reports of secondary outcomes.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Experimental (Liposomal Bupivacaine) | Control (Normal Saline)
Number analyzed (Participants) | 26 | 25
Score on a scale | 5.7 (2.2) | 6.1 (2.7)
Statistical Analysis 1: Comparison: Experimental (Liposomal Bupivacaine) vs Control (Normal Saline); Test type: Superiority; p = 0.54, t-test, 2 sided

3. Secondary Outcome: Mean NRS Pain Score at Rest on Postoperative Day 2
Description: Mean of patient-reported NRS pain scores on postoperative day 2. Patients recorded pain scores at rest with each oral analgesic tablet taken. Zero implies no pain, whereas a score of 10 translates to very severe pain. Outcome score is mean of reported pain scores for this day.
Time Frame: Postoperative day 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental (Liposomal Bupivacaine) | Control (Normal Saline)
Number analyzed (Participants) | 26 | 25
score on a scale | 5.2 (2.3) | 6.4 (2.4)
Statistical Analysis 1: Comparison: Experimental (Liposomal Bupivacaine) vs Control (Normal Saline); Test type: Superiority; p = 0.07, t-test, 2 sided

4. Secondary Outcome: Mean NRS Pain Scores at Rest on Postoperative Day 3
Description: Patients recorded their pain scores at rest with ingestion of each oral analgesic table on postoperative day 3. Zero implies no pain, whereas 10 implies very severe pain. Outcome score is mean of reported pain scores for this day.
Time Frame: Postoperative Day 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental (Liposomal Bupivacaine) | Control (Normal Saline)
Number analyzed (Participants) | 26 | 25
score on a scale | 4.6 (1.7) | 6.3 (2.2)
Statistical Analysis 1: Comparison: Experimental (Liposomal Bupivacaine) vs Control (Normal Saline); Test type: Superiority; p = 0.003, t-test, 2 sided

5. Secondary Outcome: Mean NRS Pain Score With Motion
Description: NRS Pain score with passive motion (for those patients who performed this), on 0-10 scale, with zero being no pain and 10 representing severe pain. Outcome score is mean of reported pain scores for passive motion episodes on all three postoperative days.
Time Frame: Mean value of reported pain scores on postoperative days 1,2 and 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Experimental (Liposomal Bupivacaine) | Control (Normal Saline)
Number analyzed (Participants) | 26 | 25
Score on a scale | 4.5 (3.3) | 5.1 (3.8)
Statistical Analysis 1: Comparison: Experimental (Liposomal Bupivacaine) vs Control (Normal Saline); Test type: Superiority; p = 0.53, t-test, 2 sided

6. Secondary Outcome: Oral Analgesic Requirements on Postoperative Day 1
Description: Oral analgesic dose (5 mg oxycodone tablets) required expressed as oral morphine equivalents. Outcome is total oral opioid used on postoperative day 1 expressed as oral morphine equivalents in mg.
Time Frame: Postoperative day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Oral morphine equivalents in mg
Arm/Group | Experimental (Liposomal Bupivacaine) | Control (Normal Saline)
Number analyzed (Participants) | 26 | 25
Oral morphine equivalents in mg | 42.9 (22.3) | 41.4 (29.0)
Statistical Analysis 1: Comparison: Experimental (Liposomal Bupivacaine) vs Control (Normal Saline); Test type: Superiority; p = 0.84, t-test, 2 sided

7. Secondary Outcome: Oral Analgesic Requirements on Postoperative Day 2
Description: Amount of oral opioids (oxycodone 5 mg tablets) ingested by patients on Postoperative Day 2, expressed as Oral Morphine Equivalents in mg.
Time Frame: Postoperative day 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Oral morphine equivalents in mg
Arm/Group | Experimental (Liposomal Bupivacaine) | Control (Normal Saline)
Number analyzed (Participants) | 26 | 25
Oral morphine equivalents in mg | 36.6 (30.3) | 39.0 (24.0)
Statistical Analysis 1: Comparison: Experimental (Liposomal Bupivacaine) vs Control (Normal Saline); Test type: Superiority; p = 0.76, t-test, 2 sided

8. Secondary Outcome: Oral Analgesic Requirements on Postoperative Day 3
Description: Patients reported the number of oral analgesic tablets (5 mg oxycodone tablets) ingested on postoperative day 3. This is expressed as Oral Morphine Equivalents in mg.
Time Frame: Postoperative Day 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Oral morphine equivalents in mg
Arm/Group | Experimental (Liposomal Bupivacaine) | Control (Normal Saline)
Number analyzed (Participants) | 26 | 25
Oral morphine equivalents in mg | 29.8 (34.9) | 36.4 (24.6)
Statistical Analysis 1: Comparison: Experimental (Liposomal Bupivacaine) vs Control (Normal Saline); Test type: Superiority; p = 0.44, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: The first three postoperative days.
Arm/Group | Experimental (Liposomal Bupivacaine) | Control (Normal Saline)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 18/27 | 17/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (Liposomal Bupivacaine) (N=27) | Control (Normal Saline) (N=27)
Pruritis (Skin and subcutaneous tissue disorders) | 4 | 6 — Itching. This was likely due to taking oral opioids. Solicited by questionnaire.
Nausea (Gastrointestinal disorders) | 3 | 3 — Patient complaint of nausea. Solicited by questionnaire
Insomnia (General disorders) | 7 | 10 — Patient report of difficulty with sleeping. Solicited by questionnaire
Fever (General disorders) | 2 | 0 — Patient report of increased body temperature or perception of such.Solicited by questionnaire
Headache (Nervous system disorders) | 0 | 2 — Patient complaint of pain in head. Solicited by questionnaire
Dizziness (Nervous system disorders) | 2 | 0 — Patient report of lightheadedness or vertigo-type sensation. Solicited by questionnaire
Constipation (Gastrointestinal disorders) | 9 | 6 — Patient complaint of infrequent or difficult bowel movement. Solicited by questionnaire
Poor appetite (General disorders) | 3 | 4 — Patient complaint of loss of appetite or lack of desire to eat. Solicited by questionnaire

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT03149887/Prot_SAP_000.pdf